CLINICAL TRIAL: NCT05924334
Title: Effect of Kundalini Reiki Intervention on the Symptoms of Premenstrual Syndrome and Quality of Life in Nursing Students: Randomized Controlled Trial
Brief Title: Reiki & Premenstrual Syndrome & Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Selin PAKER, Research Assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-4.1T/88
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Quality of Life
Keywords: quality of life; reiki; premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: In the research, practitioners and evaluator are different from each other. While the International Researcher with the International IAOTH -approved "Kundalini Reiki Master" certificate, he will be the Primary practitioner, one of the two other researchers will be a placebo practitioner and the other evaluator. In this way, the bias of the practitioners and the evaluation will disappear and triple blinding will be performed and reliable results will be obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reiki (Experimental): Processing steps of Reiki application; During the Reiki process, the practitioner will keep the hands just above the recipient. It will be explained to the individual that he may feel the feeling of temperature, tingling, drowsiness, refreshment or healing during therapy.
  During the application, the person does not need to be in a lying position or remove their clothes. It is enough to remove the jewelry on it.
  In order to ensure the flow of energy during the application, the arms and legs of the individual should stand open on both sides of the body, and the hands and feet will not be crossed in order not to disrupt the flow of energy.
  The practitioner will pass the right side of the individual and correct the energy existing around the body with the right hand to the feet and from top to bottom by correcting the energy field of the individual.
  The application time will be between 20 and 30 minutes on average.
  Interventions: Other: reiki
- placebo control (Experimental): The same intervention procedure will be performed with the Reiki Group. Only the placebo group practitioner does not have a Reiki Master certificate. In other words, despite the apparent reiki applied, there will be no energy flow in its real meaning.
  Interventions: Other: placebo

INTERVENTIONS:
Other: reiki — Processing steps of Reiki application; During the Reiki process, the practitioner will keep the hands just above the recipient. It will be explained to the individual that he may feel the feeling of temperature, tingling, drowsiness, refreshment or healing during therapy.
  During the application, the person does not need to be in a lying position or remove their clothes. It is enough to remove the jewelry on it.
  In order to ensure the flow of energy during the application, the arms and legs of the individual should stand open on both sides of the body, and the hands and feet will not be crossed in order not to disrupt the flow of energy.
  The practitioner will pass the right side of the individual and correct the energy existing around the body with the right hand to the feet and from top to bottom by correcting the energy field of the individual.
  The application time will be between 20 and 30 minutes on average.
  Arms: reiki
Other: placebo — placebo
  Arms: placebo control

SUMMARY:
It is planned to perform a triple blind, randomized and placebo -controlled type in order to determine the effect of Kundalini reiki application on the symptoms of premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome is common as a number of cognitive and emotional symptoms that started about a week before menstruation and has negative effects on the quality of life of women. In this period, symptoms affecting the quality of life are often listed as pain, bloating, edema, appetite changes, weight gain, tenderness, fullness, fatigue, drowsiness, anxiety, depressive symptoms and crying. It is known that women resorted to various methods that are pharmacological or non-pharmacological methods to deal with these symptoms in the premenstrual period. These methods vary from analgesic to hot application or traditional and complementary methods. Reiki is a healing energy that is not exactly included in traditional and complementary practices but has been revealed by research. In short, it is an energy therapy that balances the body and has no negative side effects. There are two types: Usui Reiki and Kundalini Reiki. From this point of view, it is planned to perform a triple blind, randomized and placebo controlled type in order to determine the effect of Kundalini reiki application on the symptoms of premenstrual syndrome. The study is planned to be carried out with Ege University Faculty of Nursing between June 2023 and July 2023. The universe of the study will consist of all students studying at the faculty in 2022-2023. The first stage of the study, which is planned to be carried out in two stages, will be made of descriptive-specific type to determine the students with premenstrual syndrome, no sample selection will not be selected and all the students who meet the criteria of inclusion in the research will be taken. In the second stage, intervention and placebo groups will be identified by randomization among students with premenstrual syndrome. In the Premenstrual periods, Reiki application will be held in the Premenstrual periods and no energy work will be applied to the placebo group. For the second stage, the adequacy of the number of samples will be decided by making power analysis during the study. Research data will be collected by face-to-face interview method using the individual promotion form, premenstrual syndrome scale and SF-36 quality of life scale and SPSS 22.0 package program will be used in statistical data analysis. At the end of the study, although the effectiveness of reiki application against premenstrual symptoms in nursing students is determined, awareness will be created to be used as a applicable method for the development of premenstrual symptom management and quality of life if the result is effective.

ELIGIBILITY:
Inclusion Criteria:

* PMS scale total score is 110 points and above
* Being a volunteer to participate in the reiki application

Exclusion Criteria:

* Having a pacemaker (Reiki application is not recommended.)
* Being pregnant (Reiki application is not recommended.)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Intensity of premenstrual symptoms evaluated using the Premenstrual Syndrome Scale | change from baseline (before implementation) and 1st week of practice
  The total score of the scale is obtained from the sum of the scores obtained from all sub -dimensions. At least 44 points can be obtained from the scale. Increased score from the scale states that the density of PMS symptoms increased
quality of life evaluated using the SF-36 Scale | change from baseline (before implementation) and 1st week of practice
  Physical function, social functionality, physical role difficulty, emotional role difficulty, energy/vitality, mental health, pain and general health perception. Subscales evaluate health between 0 and 100, and 0 shows the bad health status, while 100 good health status

CONTACTS AND LOCATIONS:
Overall Officials: Figen Kazankaya, Master, Study Chair — Ege University; Gül Ertem, PhD, Study Director — Ege University
Locations (1):
- Turkey, Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No